CLINICAL TRIAL: NCT06360354
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 193 in Combination With Other Therapies in Subjects With Advanced Gastrointestinal, Biliary Tract, or Pancreatic Cancers With Homozygous MTAP-deletion
Brief Title: A Study Evaluating AMG 193 in Combination With Other Therapies in Participants With Advanced Gastrointestinal, Biliary Tract, or Pancreatic Cancers With Homozygous Methylthioadenosine Phosphorylase (MTAP)-Deletion (MTAPESTRY 103)
Acronym: MTAPESTRY 103
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230223
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Gastrointestinal, Biliary Tract, and Pancreatic Cancers
Keywords: Advanced Cancer; Methylthioadenosine Phosphorylase; AMG 193; Oncology
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subprotocol B: Pancreatic Ductal Adenocarcinoma (PDAC) Arm A (Experimental): Part 1: Participants with MTAP-deleted PDAC will receive doses of AMG 193 orally in combination with gemcitabine and nab-paclitaxel IV.
  Part 2: Participants with MTAP-deleted PDAC will receive the recommended dose of AMG 193 in combination with gemcitabine and nab-paclitaxel.
  Interventions: Drug: AMG 193; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Subprotocol B: PDAC Arm B (Experimental): Part 1: Participants with MTAP-deleted PDAC will receive doses of AMG 193 orally in combination with mFOLFIRINOX (irinotecan, fluorouracil, leucovorin calcium, oxaliplatin) IV.
  Part 2: Participants with MTAP-deleted PDAC will receive the recommended dose of AMG 193 in combination with mFOLFIRINOX.
  Interventions: Drug: AMG 193; Drug: Modified FOLFIRINOX
- Subprotocol C: Dose Exploration (Experimental): Part 1: Participants with MTAP-deleted PDAC will receive oral doses of AMG 193 and RMC-6236.
  Interventions: Drug: AMG 193; Drug: RMC-6236
- Subprotocol C: Dose Expansion (Experimental): Part 2: Participants with MTAP-deleted PDAC will receive oral doses of AMG 193 andRMC-6236.
  Interventions: Drug: AMG 193; Drug: RMC-6236

INTERVENTIONS:
Drug: AMG 193 — Administered Orally
Drug: Gemcitabine — Administered IV
  Arms: Subprotocol B: Pancreatic Ductal Adenocarcinoma (PDAC) Arm A
Drug: Nab-paclitaxel — Administered IV
  Arms: Subprotocol B: Pancreatic Ductal Adenocarcinoma (PDAC) Arm A
Drug: Modified FOLFIRINOX — Modified FOLFIRINOX consists of irinotecan, 5-FU, LV, and oxaliplatin administered IV
  Arms: Subprotocol B: PDAC Arm B
Drug: RMC-6236 — Administered orally
  Arms: Subprotocol C: Dose Expansion; Subprotocol C: Dose Exploration

SUMMARY:
The study aims to determine maximum tolerated dose (MTD) or recommended combination dose of the MTA-cooperative PRMT5 inhibitor AMG 193 administered in combination with other therapies in adult participants with metastatic or locally advanced methylthioadenosine phosphorylase (MTAP)-deleted gastrointestinal, biliary tract, or pancreatic cancers. The study also aims to determine the safety profile of AMG 193 administered in combination with other therapies in adult participants with metastatic or locally advanced MTAP-deleted gastrointestinal, biliary tract, or pancreatic cancers.

ELIGIBILITY:
Subprotocol B

Inclusion:

* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years).
* Histologically or cytologically confirmed diagnosis of metastatic and/or unresectable (locally advanced) adenocarcinoma of the pancreas.
* Tumor tissue (FFPE sample) or an archival block must be available. Participants without archived tumor tissue available may be allowed to enroll by undergoing tumor biopsy before dosing.
* Homozygous MTAP-deletion.
* Disease measurable as defined by RECIST v1.1.
* Adequate organ function as defined in the protocol.

Exclusion:

* Prior treatment with a MAT2A inhibitor or a PRMT5 inhibitor.
* Radiation therapy within 28 days of first dose.
* Major surgery within 28 days of first dose of AMG 193.
* Cardiovascular and pulmonary exclusion criteria as defined in the protocol.
* Gastrointestinal tract disease causing the inability to take PO medication, malabsorption syndrome, requirement for IV alimentation, gastric/jejunal tube feeds, uncontrolled inflammatory gastrointestinal disease (eg, Crohn's disease, ulcerative colitis).
* History of solid organ transplantation.

Subprotocol C

Inclusion:

* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years).
* Histologically or cytologically confirmed diagnosis of metastatic and/or unresectable (locally advanced) adenocarcinoma of the pancreas.
* Homozygous MTAP-deletion.
* Rat Sarcoma Viral Oncogene Homolog (RAS) mutation
* Received at least 1 prior systemic therapy for advanced or metastatic PDAC.
* Disease measurable as defined by RECIST v1.1.
* Adequate organ function as defined in the protocol.

Exclusion:

* Prior treatment with aMAT2A inhibitor, a PRMT5 inhibitor, or a MAPK pathway inhibitor, including KRAS inhibitors.
* Cardiovascular and pulmonary exclusion criteria as defined in the protocol.
* Gastrointestinal tract disease causing the inability to take PO medication, malabsorption syndrome, requirement for IV alimentation, gastric/jejunal tube feeds, uncontrolled inflammatory gastrointestinal disease (eg, Crohn's disease, ulcerative colitis).
* History of solid organ transplantation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2029-02-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose Limiting Toxicities (DLT) | Up to 28 days
Number of Participants Experiencing Treatment Emergent Adverse Events (TEAE) | Up to approximately 2 years
  Any clinically significant changes in vital signs, electrocardiogram, or lab parameters will be recorded as TEAEs.
Number of Participants Experiencing Serious Adverse Events (SAE) | Up to approximately 2 years

SECONDARY OUTCOMES:
Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to approximately 2 years
Disease Control (DC) per RECIST v1.1 | Up to approximately 2 years
Duration of Response (DOR) per RECIST v1.1 | Up to approximately 2 years
Time to Response (TTR) per RECIST v1.1 | Up to approximately 2 years
Overall Survival (OS) per RECIST v1.1 | Up to approximately 2 years
Progression-free Survival (PFS) per RECIST v1.1 | Up to approximately 2 years
Maximum Plasma Concentration (Cmax) of AMG193 | Up to Day 1 of Cycle 5 (one cycle = 21 or 28 days)
Time to Maximum Plasma Concentration (tmax) of AMG193 | Up to Day 1 of Cycle 5 (one cycle = 21 or 28 days)
Area Under the Plasma Concentration-time Curve (AUC) of AMG 193 | Up to Day 1 of Cycle 5 (one cycle = 21 or 28 days)
Cmax of RMC-6236 | Up to Day 1 of Cycle 5 (one cycle = 21 days)
Tmax of RMC-6236 | Up to Day 1 of Cycle 5 (one cycle = 21 days)
AUC of RMC-6236 | Up to Day 1 of Cycle 5 (one cycle = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (77):
- United States (29):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Translational Research in Oncology US Inc, Trio Central Pharmacy, Los Angeles, California
  - University of California Los Angeles, Santa Monica, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - Oncology Consultants Cancer Center, Houston, Texas
  - US Oncology Research Investigational Products Center, Irving, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialists PC, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
- Australia (6):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - GenesisCare -North Shore Oncology, St Leonards, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Austin Health, Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth Healthcare, St Albans, Victoria
- Belgium (3):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Canada (3):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHU de Quebec Hopital de l Enfant Jesus, Québec, Quebec
- China (6):
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
- Herlev og Gentofte Hospital, Herlev, Denmark
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Institut Paoli Calmettes, Marseille
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - Alexandra Hospital, Athens
  - General Hospital Of Thessaloniki Papageorgiou, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Centro Ricerche Cliniche Di Verona Societa responsabilita limitata, Verona
- Japan (4):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Spain (3):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital General Universitario Gregorio Maranon, Madrid
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Sarah Cannon Research Institute UK, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com